CLINICAL TRIAL: NCT04998591
Title: Effects of Fasting on Success Rates of In-vitro-fertilization (IVF) / Intracytoplasmatic Sperm Injection (ICSI) in Women With Fertility Disorders
Brief Title: Effects of Fasting on Success Rates of Assisted Reproductive Techologies
Acronym: KiWuC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KiWuC
Record Dates: First submitted 2021-07-24; First posted 2021-08-10 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Sub Fertility, Female; Fertility Disorders; Fertility Issues; Sub-fertility; IVF
Keywords: fasting; natural therapies; caloric restriction; lifestyle modification; dietary restriction; dietary intervention; complementary medicine; integrative medicine; Intracytoplasmatic sperm injection ICSI
MeSH Terms: conditions — Infertility, Female; Infertility; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: This explorative study is conducted in form of a randomized, controlled trial design with a fasting intervention and a waiting list, which continues the usual diet.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask a fasting intervention for the participant or the study personel. Therefore only outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (Experimental): Participants will be councelled and accompanied to follow a fasting regime of 7 days in an outpatient setting under medical supervision.
  Interventions: Behavioral: Fasting
- Waiting list (No Intervention): This group maintains their individual diet during the whole time of the study. In case that the first cycle of In-Vitro-Fertilization fails, they are offered a fasting intervention before a next cycle.

INTERVENTIONS:
Behavioral: Fasting — fasting for 7 days (caloric intake <500 kcal in liquid form)
  Other Names: Prolonged Fasting
  Arms: Fasting group

SUMMARY:
This exploratory study investigates fasting as a potential supportive therapy for infertility treatment in women undergoing in-vitro-fertilization (IVF) / intracystoplamsatic sperm injection (ICSI)

DETAILED DESCRIPTION:
This 2-arm, randomized, controlled exploratory clinical trial aims to explore fasting as a novel supportive treatment in female infertility during IVF / ICSI. The participants will be randomized in two groups: a fasting group and a waiting list. The intervention group follows a fasting intervention, whereas the patients on the waiting list continue their normal diet. All groups will be trained and accompanied by medical experts. In addition, qualitative interviews will be conducted including individual and focus group interviews with a subgroup of participants.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 to 38 years with planned IVF / ICSI
* 1 ng/ml ≤ Anti-Mullerian Hormone (AMH) ≤ 4 ng/ml
* Unfulfilled desire to have children >1 year
* 25 kg/m² ≤ BMI ≤ 35 kg/m² declaration of consent

Exclusion Criteria:

* Language barriers
* Previously known serious mental illness or cognitive impairment
* Patients with anatomical/organic damage and proven uterine abnormalities
* Eating disorders in the medical history
* Serious previous internal diseases
* Lack of internet access
* No consent to randomisation
* Participation in other studies

Ages: 25 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biological female sex
Enrollment: 1 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Fertilisation rate | throughout 1-3 days after in-vitro-fertilization (IVF) / intracytoplasmatic sperm injection (ICSI)
  Fertilisation rate of the retrieved oocytes

SECONDARY OUTCOMES:
glucose in culture medium of oocytes | throughout 1-3 days after in vitro fertilisation
  chemical composition of culture medium (glucose)
lactate in culture medium of oocytes | throughout 1-3 days after in vitro fertilisation
  chemical composition of culture medium (lactate)
pyruvate in culture medium of oocytes | throughout 1-3 days after in vitro fertilisation
  chemical composition of culture medium (pyruvate)
pregnancy rate | 4 weeks after IVF/ICSI
  pregnancies after IVF/ICSI
rate of mature oocytes | at IVF / ICSI intervention
  rate of mature oocytes
rate of life births | 10 months after IVF/ICSI
  rate of life births after IVF/ICSI
rate of implantable embryos | at IVF/ICSI
  rate of implantable embryos after the IVF/ICSI
Course of IVF/ICSI preparation and pregnancy | 4 weeks and 10 months after IVF / ICSI
  Course of IVF/ICSI preparation and pregnancy
WHO-5 questionnaire | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  Quality of life
changes in diet | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  self-developed questionnaire to examine dietary behaviour
mindfulness | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  MAAS-questionnaire, validated questionnaire to examine mindfulness
anxiety and depression | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  HADS-questionnaire, validated questionnaire to examine anxiety and depression
current mood | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  ASTS-questionnaire, validated questionnaire to examine current mood
experienced stress | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  Cohen-stress scale, validated questionnaire to examine experienced stress
physical fitness | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  questionnaire to examine physical fitness
quality of relationship | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  self-developed questionnaire to examine the relationship between the two partners desiring to have a child
psychological stress caused by the unfulfilled desire to have children | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  self-developed questionnaire to examine the psychological stress caused by the unfulfilled desire to have children
gratitude | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  validated questionnaire to examine gratitude
self-efficacy | baseline, within one week before IVF, 4 weeks after IVF, 10 months after baseline
  ASKU, validated questionnaire to examine self-efficacy
abdominal sonography | within 1 month before, during and within 2 weeks after the fasting intervention
  sonography in a subgroup

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Hochschulambulanz für Naturheilkunde der Charité-Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: after the end of the study for 5 years
Access Criteria: on demand